CLINICAL TRIAL: NCT03623217
Title: Development and Validation of the Questionnaire in Assessing the Health-related Quality of Life of Patients Who Switch From b.i.d to q.d of Tacrolimus After Kidney Transplantation
Brief Title: Quality of Life Questionnaire Validation for Patients With Changed Tacrolimus Dosing After Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: ADV-KT-14-01
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2018-10

CONDITIONS: Kidney Transplantation
Keywords: Behavioral; Questionnaire development; Questionnaire; Interview with patients; Observational; Tacrolimus; Patient reported outcome tool; Validation; Kidney transplantation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant participants receiving tacrolimus: Transplant participants who have received tacrolimus twice daily for a minimum of 6 months to a maximum of 12 months after the surgery, and who are within 1 month of switching to the once daily regimen of modified release tacrolimus.
  Interventions: Behavioral: Qualitative interviews with participants

INTERVENTIONS:
Behavioral: Qualitative interviews with participants — For the development and validation of a questionnaire.

SUMMARY:
The purpose of this study is to develop and validate a questionnaire to assess the quality of life when the recipients of kidney transplantation switched their medication from tacrolimus twice daily (BID regimen) to Advagraf (once daily (QD) regimen of modified release tacrolimus).

DETAILED DESCRIPTION:
This study will develop and validate a questionnaire to assess the health-related quality of life when switching from tacrolimus twice daily (b.i.d) regimen to once daily (q.d) regimen after kidney transplantation.

In-depth interviews are conducted to develop questionnaire items, and the interviewees are as follows: participants who have received tacrolimus b.i.d for a minimum of 6 months to a maximum of 12 months, and who are within 1 month of switching to Advagraf (q.d regimen of modified release tacrolimus).

The time required for the in-depth interview is approximately 30 minutes to one hour.

After questionnaire items are developed, survey participants for validation are as follows: the first survey is conducted on participants who have received tacrolimus b.i.d for a minimum of 6 months to a maximum of 12 months during the period. The second survey is conducted within one month after switching to Advagraf (q.d regimen of modified release tacrolimus).

At the validation stage, the survey using the developed questionnaire is conducted twice, once during the b.i.d. regimen and once after switching to the q.d. regimen.

ELIGIBILITY:
Inclusion Criteria

Selection criteria for in-depth interview subjects:

* One male or female aged 30 or over but below 40 years old.
* One male or female aged 60 or over but below 70 years old.
* One male or female with an occupation.
* One male or female without an occupation.
* Two subjects, depending on the number of medications (more or less medications) that the subject is taking.
* Participation available Period: subjects who have received tacrolimus twice daily (b.i.d) for a minimum of 6 months to a maximum of 12 months after surgery and who are within 1 month of switching to Advagraf (once daily (q.d) regimen of modified release tacrolimus).
* Subjects who understood the purpose and risks of the questionnaire development and who were well-acquainted with the contents and submitted the written consent to participate in the interview for the questionnaire development.

Selection criteria for validation stage subjects:

1. Males and females aged 19 to 65 years old.
2. Participation Available Period: the first survey is conducted on the subjects who have received tacrolimus twice daily (b.i.d) for a minimum of 6 months to a maximum of 12 months during the period. The second survey is conducted within one month after switching to Advagraf (once daily (q.d) regimen of modified release tacrolimus).
3. Subjects who understood the purpose and risks of the questionnaire development and who were well-acquainted with the contents and submitted the written consent to participate in the interview for the questionnaire development.

Exclusion Criteria:

* None.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who underwent kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life(HRQoL) measured by the newly developed and validated Kidney Transplantation and Quality of Life(KTQoL) Questionnaire | Up to a maximum of 32 months
  KTQoL is a transplantation-specific questionnaire to assess 'General QoL' for transplant participants after surgery and 'Specific QoL' for transplant participants after conversion from twice-daily (BID) to once-daily (QD) tacrolimus. 'General QoL' represents how good the participant's HRQoL is after a transplant surgery and 'Specific QoL' shows how good the participant's health is after conversion of medication from BID to QD. The KTQoL questionnaire consists of 24 questions, 17 for 'General Health' and 7 for 'Specific Health'. The total 'General QoL' scores range from 0-58 and it has sub-scales scores of global scale (range of 0-4), worry (range of 0-16), symptom (range of 0-28) and everyday life (range of 0-10). The total 'Specific QoL' scores range from 0-22 with no sub-scales. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Pharma Korea, Inc., Study Chair — Astellas Pharma Korea, Inc.
Locations (1):
- Site 1, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.